CLINICAL TRIAL: NCT06491004
Title: Evaluation of DiaSorin LIAISON® PTX3 (Long Pentraxin 3) Assay in Patients With Pneumonia
Status: Completed | Type: Observational
Sponsor: Diasorin Italia S.p.A. (Industry)
Responsible Party: Sponsor
Other Study IDs: CLI-PR-2104
Record Dates: First submitted 2024-06-06; First posted 2024-07-08 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-07

CONDITIONS: Pneumonia
MeSH Terms: conditions — Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — After collection, plasma and urine samples will be immediately processed, coded, and stored frozen at <- 20 °C.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: PTX3 assay — PTX3 dosage by the in vitro medical device in evaluation.

SUMMARY:
LIAISON® PTX3 is an in vitro chemiluminescent immunoassay (CLIA) intended for the quantitative determination of Long Pentraxin 3 (PTX3) in human plasma samples.

LIAISON® PTX3, in conjunction with clinical evaluation and other laboratory findings, may serve as an aid in the determination of disease severity and prognosis of patients with community-acquired (CAP) and hospital-acquired pneumonia (HAP), including ventilator-associated pneumonia (VAP).

DETAILED DESCRIPTION:
Long Pentraxin 3 (PTX3) is an essential protein of innate immunity, produced by myeloid cells, endothelial cells and respiratory epithelial cells, and involved in resistance to selected pathogens and in inflammation. In different pathological conditions (infections of bacterial and viral origin, sepsis, and cardiovascular diseases) and in patients requiring admission to intensive care units (ICUs), PTX3 was detected in high concentrations in the circulation and was associated with disease severity and mortality.

PTX3 plasma concentration was found to be an independent prognostic indicator of short-term mortality (28 days) in hospitalized patients with Coronavirus Disease 2019 (COVID- 19) and higher PTX3 levels were found in ICU patients compared to ward patients. Moreover, PTX3 significantly correlated with the inflammatory molecules C-reactive protein (CRP), procalcitonin (PCT), and interleukin (IL)-6.

Given the association between PTX3 and inflammatory conditions, especially in the context of lung infections, the study aims to investigate the potential of PTX3 to be used as a severity marker and a prognostic predictor for outcome in patients with community-acquired (CAP) and hospital-acquired pneumonia (HAP), including ventilator-associated pneumonia (VAP).

ELIGIBILITY:
Inclusion Criteria:

* Subjects willing and able to sign the approved Informed Consent form in accordance with international and national regulations
* Patients diagnosed with pneumonia, either CAP, HAP, VAP
* Collection of plasma samples within 24 hours from pneumonia diagnosis (for CAP diagnosis is usually made at ED presentation and for HAP and VAP diagnosis is made during hospital stay)
* K2 EDTA plasma samples dedicated to the study have a minimum volume of 3 mL

Exclusion Criteria:

* Patients who are currently pregnant
* Samples collected and/or stored in an inappropriate way

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with either CAP, HAP or VAP. Based on clinical evaluation and pneumonia severity assessment, patients will be hospitalized (in-patients) or not hospitalized (out-patients).
Sampling Method: Non-Probability Sample
Enrollment: 281 (Actual)
Dates: Start 2021-09-20 (Actual); Primary Completion 2024-03-29 (Actual); Study Completion 2024-03-29 (Actual)

PRIMARY OUTCOMES:
Pneumonia severity measured by pneumonia specific index (PSI), CURB-65, and Sequential Organ Failure Assessment (SOFA) as a mortality prediction score | Day 0 (baseline), day 3, day 7, at discarge, an average of 1 month (if applicable)
  Evaluate Long Pentraxin 3 (PTX3) correlation with pneumonia severity and clinical outcome: pneumonia severity is assessed by clinical scores, specifically pneumonia severity index (PSI), CURB-65, Sequential Organ Failure Assessment (SOFA) and Horowitz Index as a mortality prediction score; clinical outcome means hospitalization, intensive care unit (ICU) admission, mortality (at 28 days), discharge.
  PSI (pneumonia severity) score: I or II MILD; III MODERATE; IV or V SEVERE. CURB-65 score: 0-1 MILD; 2 MODERATE; 3-4-5 SEVERE SOFA score: 0 to 3 MILD; 4 to 9 MODERATE; 10 to 14 or more SEVERE
  Clinical severity:
  presence of unilateral pneumonia with less than 50% parenchymal involvement; basal bilateral pneumonia LOW unilateral pneumonia with more than 50% parenchymal involvement; bilateral with involvement of a large area of parenchyma HIGH
  Horowitz Index (P/F ratio), mmHg:
  >300 no distress respiratory syndrome; >200 to 300 MILD; >100 to 200 MODERATE; <=100 SEVERE
PTX3 cutoffs | Day 0 (baseline), day 3, day 7, at discarge, an average of 1 month (if applicable)
  Identify PTX3 cutoffs (LIAISON® PTX3 assay) to distinguish pneumonia severity: pneumonia severity is assessed by clinical scores (PSI, CURB-65, SOFA and Horowitz Indexas a mortality prediction score).
  Details in Primary Outcome Measure 1

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Istituto Clinico Humanitas, Rozzano, Milan
  - Cliniche Humanitas Gavazzeni, Bergamo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Voza A, Aliberti S, Bonelli F, Ingallinella P, Ghezzi E, Mauro C, Rossini C, Mastronardo C, Felotti S, Bottazzi B, Garlanda C, Zierold C, Ghignoni G, Mantovani A. A machine learning model including pentraxin-3 as predictor of outcomes in community-acquired pneumonia. J Transl Med. 2025 Oct 31;23(1):1205. doi: 10.1186/s12967-025-07142-6. PMID 41174667